CLINICAL TRIAL: NCT02470871
Title: Multi-center, Randomized, Open-label, Parallel-Arm, Single-dose, Pharmacokinetic Study of rVIIa-FP (CSL689) in Subjects With Congenital Factor VII Deficiency
Brief Title: Study of the Pharmacokinetics and Safety of Recombinant Factor VIIa Fusion Protein (rVIIa-FP, CSL689) in Patients With Congenital Factor VII Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSL689_1002; 2014-002982-32 (EudraCT Number)
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-11

CONDITIONS: Congenital Coagulation Factor VII Deficiency
MeSH Terms: interventions — recombinant FVIIa

ARMS (2):
- Low-dose CSL689 (Experimental): Single dose of subject's routine FVII replacement therapy (either eptacog alfa [activated] [ie, comparator drug 1] or pdFVII [ie, comparator drug 2]), followed by a single dose of CSL689 at the low dose
  Interventions: Biological: Eptacog alfa (activated) or pdFVII; Biological: CSL689
- High-dose CSL689 (Experimental): Single dose of subject's routine FVII replacement therapy (either eptacog alfa [activated] [ie, comparator drug 1] or pdFVII [ie, comparator drug 2]), followed by a single dose of CSL689 at the high dose.
  Interventions: Biological: Eptacog alfa (activated) or pdFVII; Biological: CSL689

INTERVENTIONS:
Biological: Eptacog alfa (activated) or pdFVII — Comparator Drug 1: Recombinant activated FVII (rFVIIa). Subjects with eptacog alfa (activated) as their routine FVII replacement therapy will receive a single dose of eptacog alfa (activated) in the study.
  Comparator Drug 2: Plasma-derived FVII (pdFVII). Subjects with pdFVII as their routine FVII replacement therapy will receive a single injection of pdFVII in the study.
Biological: CSL689 — Experimental Drug: Recombinant fusion protein, linking activated FVII with albumin (rVIIa-FP). Subjects will receive a single dose of CSL689 at either a low dose (Arm 1) or a high dose (Arm 2)

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics (PK) and safety of rVIIa-FP (CSL689) in a total of 10 to 16 male or female adults with inherited coagulation factor VII (FVII) deficiency. Subjects will receive a single dose of their routine FVII replacement product (ie, either recombinant activated coagulation FVII [rFVIIa, eptacog alfa (activated)] or plasma-derived FVII [pdFVII]) as a comparator, and will then be randomly assigned to a single low dose or a single high dose of the study product CSL689 (8 subjects per CSL689 dose level). Serial blood samples for PK analysis will be taken up to 24 hours after the eptacog alfa (activated) or pdFVII injection, and up to 48 hours after the CSL689 injection. Subject safety will be routinely monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Proven congenital FVII deficiency.
* Age ≥ 18 years.
* FVII level < 2% of normal levels.
* Minimum of 50 previous exposure days to pdFVII (including prothrombin complex concentrates [PCCs]) or rFVIIa.

Exclusion Criteria:

* History of, or risk factors for, thromboembolic events, including known deep vein thrombosis.
* Inhibitor to FVII or rFVIIa, current or historic.
* Known or suspected hypersensitivity to hamster protein, to CSL689, or to any excipient of CSL689.
* Known or suspected allergy to rFVIIa or hamster protein.
* Major surgery within 1 month before screening.
* Advanced atherosclerotic disease (ie, known history of ischemic heart disease, or ischemic stroke).
* Human immunodeficiency virus (HIV)-positive subjects with cluster of differentiation 4 (CD4)+ lymphocyte count of < 200/µL at screening.
* Use of an investigational agent within 30 days before the study.
* Use of concomitant therapy not permitted during the study (ie, other platelet inhibitors, desmopressin, fibrinolysis inhibitors, except if used as local treatment [eg, for oral bleeds])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Terminal half-life of plasma FVIIa activity | Up to 48 hours after CSL689 injection
Maximum observed plasma FVIIa activity | Before injection and at up to 9 time points until 48 hours after injection
Area under the curve (AUC0-t) | Before injection and at up to 9 time points until 48 hours after injection
  Area under plasma FVIIa activity versus time curve from time 0 to last sample with quantifiable activity

SECONDARY OUTCOMES:
Total clearance | Before injection and at up to 9 time points until 48 hours after injection
  Total clearance of plasma FVIIa activity
Volume of distribution of the terminal phase | Before injection and at up to 9 time points until 48 hours after injection
AUC(0-inf) | Before injection and at up to 9 time points until 48 hours after injection
  Area under plasma FVIIa activity versus time curve from time 0 extrapolated to infinity
Incremental recovery | Before injection and at up to 9 time points until 48 hours after injection
  Incremental recovery of plasma FVIIa activity
Time of occurrence of maximum observed plasma FVIIa activity | Before injection and at up to 9 time points until 48 hours after injection
Number of subjects with antibodies against Chinese hamster ovary protein and FVII | Up to 30 days after CSL689 injection
Number of subjects with inhibitors against FVII | Up to 30 days after CSL689 injection

CONTACTS AND LOCATIONS:
Overall Officials: Alex Veldman, Study Director — CSL Behring
Locations (2):
- Site Reference 5280023, Njmegen, Netherlands
- Site Reference # 5780001, Oslo, Norway